CLINICAL TRIAL: NCT02449395
Title: A Cross-sectional Study of Fibromyalgia in Beijing
Brief Title: Cross-sectional Study of Fibromyalgia
Status: Completed | Type: Observational
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Juan Jiao, attending physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Other Study IDs: 39301
Record Dates: First submitted 2015-05-02; First posted 2015-05-20 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is designed to collect data on precipitating factors, diagnosis, morbidity, therapy, quality of life, and symptom severity, etc. informations in patients with fibromyalgia.

DETAILED DESCRIPTION:
Patients fulfilling 1990 ACR criterion for fibromyalgia will be recruited in Fibromyalgia outpatient service which is belonged to the Department of Rheumatism. Except collecting patients' demographic and social characteristic informations, rheumatologist also carry out a comprehensive evaluation including patient current history, current medication use, and tender point examination for a diagnosis or confirmation of fibromyalgia and treatment recommendations. Patients with fibromyalgia will be asked to fill a set of questionnaires to evaluate their quality of life, symptoms severity, quality of sleep and emotion. The study will be conducted in Beijing, China.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Fulfills the American College of Rheumatology (ACR) 1990 classification criteria for Fibromyalgia.

Exclusion Criteria:

* Don't fulfill any classification criterions for Fibromyalgia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients fulfilling 1990 ACR criterion for fibromyalgia be seen in the Fibromyalgia Outpatient Service which belonged to the Department of Rheumatism, Guang'anmen Hospital, Beijing China.
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia symptoms severity as measured by Fibromyalgia Impact Questionnaire (FIQ) | up to 1 week

SECONDARY OUTCOMES:
QOL as measured by Short Form-36 Health Status Questionnaire (SF-36) | up to 1 week
Pain scores as measured by Numerical rating scale (NRS) | up to 1 week
Fatigue scores as measured by Multidimensional Assessment Fatigue (MAF) | up to 1 week
Depression scores as measured by Beck depression inventory (BDI) | up to 1 week
Stress scores as measured by Perceived Stress Scale (PSS) | up to 1 week
Sleep scores as measured by Pittsburgh sleep quality index (PSQI) | up to 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Juan Jiao, M.D.,PhD, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang Y, Liu P, Li Z, Wu S, Long M, Li Y, Jiao J, Xie Z. Quality of life, pain, depression, fatigue and sleep in patients with remission or mild fibromyalgia: a comparison with remission or low disease activity rheumatoid arthritis and healthy controls. BMC Musculoskelet Disord. 2025 Jan 18;26(1):67. doi: 10.1186/s12891-025-08323-6. PMID 39827119